CLINICAL TRIAL: NCT00023894
Title: A Phase II Evaluation of Flavopiridol (NSC# 649890) in the Treatment of Recurrent or Persistent Endometrial Carcinoma
Brief Title: Flavopiridol in Treating Patients With Recurrent or Persistent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068874; GOG-0129M
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2004-05

CONDITIONS: Endometrial Cancer
Keywords: recurrent endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — alvocidib

INTERVENTIONS:
Drug: alvocidib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of flavopiridol in treating patients who have recurrent or persistent endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of flavopiridol in patients with recurrent or persistent endometrial carcinoma.
* Determine the nature and degree of toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive flavopiridol IV over 1 hour on days 1-3. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 19-51 patients will be accrued for this study within 10-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary endometrial carcinoma

  * Recurrent or persistent disease
  * Refractory to curative therapy or established treatment
* Previously treated with only 1 prior cytotoxic chemotherapy regimen (either single agent or combination therapy) for endometrial carcinoma

  * Initial treatment may include high-dose, consolidation, or extended therapy administered after surgical or non-surgical assessment
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
  * At least 1 target lesion outside previously irradiated field
* Ineligible for higher priority Gynecologic Oncology Group (GOG) protocol, defined as any active GOG phase III protocol for the same patient population

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* PT/PTT normal

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No prior thromboembolic events or thrombophlebitis
* No prior recent myocardial infarction
* No prior angina
* No prior cerebrovascular accident
* No prior transient ischemic attacks

Other:

* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No grade 2 or greater sensory or motor neuropathy
* No active infection requiring antibiotics

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic or immunologic agents for endometrial carcinoma

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy for endometrial carcinoma and recovered

Endocrine therapy:

* At least 1 week since prior hormonal therapy for endometrial carcinoma
* Concurrent hormone replacement therapy allowed

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy for endometrial carcinoma and recovered

Surgery:

* At least 3 weeks since prior surgery for endometrial carcinoma and recovered
* At least 6 months since prior re-vascularization procedures (e.g., coronary artery bypass graft, carotid endarterectomy or bypass, or angioplasty with or without stents)

Other:

* At least 3 weeks since other prior therapy for endometrial carcinoma
* At least 6 months since prior thrombolytic procedures
* No prior cyclin-dependent kinase inhibitors
* No prior anticancer therapy that would preclude study
* No concurrent amifostine or other protective reagents

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-07; Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward C. Grendys, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (54):
- United States (50):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Tuft-New England Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Barrett Cancer Center, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - CCOP - M.D. Anderson Research Base, Houston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Fletcher Allen Health Care - Medical Center Campus, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- Australia New Zealand Gynaecological Oncology Trials Group, Camperdown, New South Wales, Australia
- Tom Baker Cancer Center - Calgary, Calgary, Alberta, Canada
- Norwegian Radium Hospital, Oslo, Norway
- University of Birmingham, Birmingham, England, United Kingdom

REFERENCES:
- [Result] Grendys EC Jr, Blessing JA, Burger R, Hoffman J. A phase II evaluation of flavopiridol as second-line chemotherapy of endometrial carcinoma: a Gynecologic Oncology Group study. Gynecol Oncol. 2005 Aug;98(2):249-53. doi: 10.1016/j.ygyno.2005.05.017. PMID 15978659